CLINICAL TRIAL: NCT00691509
Title: The Role of Diet, Complementary Treatment and Lifestyle in Breast Cancer Survival
Brief Title: Dietary Phytoestrogens, Complementary and Alternative Medicine, and Lifestyle in Predicting Survival of Women With Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College London Hospitals (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000589004; UCLH-BCRG-DIETCOMPLYF-1456; EU-20823
Record Dates: First submitted 2008-06-04; First posted 2008-06-05 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2008-06

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gene Expression Profiling; Amplified Fragment Length Polymorphism Analysis; Chromatography, High Pressure Liquid; Mass Spectrometry

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: polymorphism analysis
Other: high performance liquid chromatography
Other: laboratory biomarker analysis
Other: mass spectrometry
Other: questionnaire administration

SUMMARY:
RATIONALE: Eating a diet rich in phytoestrogens may slow the growth of breast cancer cells and prevent further tumor progression. Learning about the lifestyles of women with breast cancer, their intake of phytoestrogens derived from food and supplements, and their use of complementary or alternative medicine (CAM) practices may help doctors learn more about breast cancer.

PURPOSE: This clinical trial is studying the effect of dietary and supplemental phytoestrogens and CAM therapies in preventing progression and improving survival of women with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if phytoestrogen intake affects breast cancer progression and survival in women with breast cancer.
* To consider the influence of other phytochemicals on breast cancer progression in these patients, using samples of patient blood and urine and patient-derived data.
* To develop a database of food, dietary supplements, and phytoestrogens based on data derived from these patients.
* To consider influences of diet and dietary supplements on quality of life of these patients.
* To measure 17 phytoestrogens in blood and urine samples from these patients.

OUTLINE: This is a multicenter study.

Patients undergo blood and urine sample collection once a year for 5 years during routine clinical follow-up after breast cancer diagnosis and treatment. Blood samples are frozen for future analysis of body hormones, tumor markers, and immune reactions, as well as vitamins and plant chemicals reflecting patient diet and supplements. Blood samples are also analyzed for genetic studies of cancer risk factors and polymorphisms. Urine samples are analyzed for the presence of phytoestrogens and their metabolites by immunoassays, high performance liquid chromatography (HPLC), and mass spectrometry. Some samples are analyzed for estrogenic potency by the estrogen receptor-mediated chemical activated luciferase gene expression test to assess total plasma levels of estrogen-mimics not previously detected by the other tests. Phytochemicals are also assessed.

Patients also complete a series of questionnaires once each year for 5 years and an EPIC 7-day Food Diary in years 2 and 4 to assess the role of diet and lifestyle in breast cancer survival. The questionnaires include the EORTC Quality of Life-30 to assess lifestyle; the General Health Questionnaire 12 to assess general health and levels of anxiety; and up to two Food Frequency questionnaires to assess habitual dietary intake of phytoestrogens. Patients are also asked about their use of dietary supplements and complementary and alternative medicine.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive primary breast cancer

  * Grade I to III disease
  * No bilateral disease
* Completed active treatment for primary breast cancer within 9 months to 15 months after diagnosis
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* No prior cancer except basal cell carcinoma
* No other concurrent primary cancer
* No cognitive impairment
* No psychological problems (e.g., severe endogenous depression)
* Able to understand English well

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2300 (Estimated)
Dates: Start 2005-01; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Leathem, MD, Principal Investigator — University College London Hospitals
Locations (1):
- University College Hospital, London, England, United Kingdom